CLINICAL TRIAL: NCT00271362
Title: Bone Physiology & Mechanics in Osteomyoplasty Amputation Rehabilitation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This project is no longer active with DVA.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O3789-I
Record Dates: First submitted 2005-12-28; First posted 2005-12-30 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Amputation; Fracture; Inflammation; Osteoporosis
Keywords: Exercise; Physical function; Prosthetic mobility; Rehabilitation
MeSH Terms: conditions — Fractures, Bone; Inflammation; Osteoporosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): comparing 2 surgical procedures
  Interventions: Behavioral: Amputation rehabilitation exercise program; Procedure: Osteomyoplasty vs. routine long posterior flap

INTERVENTIONS:
Behavioral: Amputation rehabilitation exercise program — participants will be physically exercised with a full array of exercise methodologies.
Procedure: Osteomyoplasty vs. routine long posterior flap — participants enrolled randomly in one of two surgical procedures.

SUMMARY:
The purpose of the study is to compare the effect of different lower limb amputation surgical procedures on leg bone integrity and rehabilitation outcome.

DETAILED DESCRIPTION:
Osteoporosis leading to increased risk of fracture, especially in the ipsilateral limb, is well documented in lower limb amputees. The purpose of this research is to examine the clinical utility of two amputation surgical procedures in: a) minimizing short and longer-term deleterious effects of amputation on bone integrity relative to the antecedents of osteoporotic change: reduced weight bearing capacity, inflammation, impaired muscle viability, and vascular compromise, and b) deriving benefit from prosthetic rehabilitation and exercise interventions.

In a randomized controlled clinical trial, we will test the hypotheses: In lower limb traumatic and dysvascular amputation, when compared to the transtibial long posterior flap amputation technique and the transfemoral Gottschalk method, the osteomyoplastic reconstruction technique developed by Ertl:

1. Hypothesis 1: results in fewer detrimental effects on bone metabolism, structure, and mass.
2. Hypothesis 2: leads to optimal rehabilitation and functional outcomes. Specifically, we will examine, in traumatic and dysvascular lower limb amputees randomly assigned to undergo either the long posterior flap amputation method or amputation with osteomyoplastic reconstruction in transtibial amputation and either the Gottschalk amputation method or amputation with osteomyoplastic reconstruction in transfemoral amputation, differences in the following parameters at baseline, 6 weeks (post-operative recuperation), and 6 months (termination of supervised rehabilitation and exercise intervention).

We will assess bone integrity in patients undergoing standard amputation versus osteomyoplastic reconstruction by measuring bone metabolism and bone mineral density and mineral content. Second, we will measure inflammatory response in patients undergoing standard amputation versus osteomyoplastic reconstruction by assessing weight bearing and impact, muscle integrity, and limb vascularity. Last, we will compare rehabilitation and functional outcome in patients undergoing standard amputation versus osteomyoplastic reconstruction by assessing prosthetic mobility, functional capacity, activity levels, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Adult lower limb PVD-related or traumatic amputees who are appropriate candidates for amputation rehabilitation exercise.

Exclusion Criteria:

1. Cognitive dysfunction (MiniMental scores <23), advanced neuropathies, or neurological impairment (CVA, Parkinson's) with residual loss of function enough to preclude exercise;
2. Unresolved MI (high isoenzymes), angina, arrhythmia, 3rd degree AV block, fixed-rate pacer;
3. Recent embolus/thrombophlebitis, myocarditis, pericarditis, or cardiomyopathy;
4. Resting SBP >200mmHg or DBP >100mmHg;
5. Uncontrolled metabolic disease, liver or kidney failure, alcohol/drug addiction; acute infection;
6. Exercise-exacerbated neuromuscular/musculoskeletal disorders; irreducible hip/leg contractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2006-01 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Bone Integrity | 6 weeks - 6 months

SECONDARY OUTCOMES:
Inflammatory Response | 6 weeks - 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Brackett, MD, Principal Investigator — VA Medical Center, Oklahoma City
Locations (1):
- VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma, United States